CLINICAL TRIAL: NCT03018483
Title: Comparison Between Automated Pressure Support Ventilation, Variable Pressure Support Ventilation and Non-variable Pressure Support Ventilation in Weaning From Mechanical Ventilation
Brief Title: Mechanical Ventilation- Weaning and Thoracic Impedance Tomography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Maria Vargas, Resercher, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSWEAN and EIT
Record Dates: First submitted 2017-01-04; First posted 2017-01-12 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Weaning From Mechanical Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Variable PSV (Experimental)
  Interventions: Device: Variable PSV
- Conventional PSV (Active Comparator)
  Interventions: Device: Conventional PSV
- Automated PSV (Active Comparator)
  Interventions: Device: Automated PSV
- NAVA (Active Comparator)
  Interventions: Device: NAVA

INTERVENTIONS:
Device: Variable PSV — Pressure support is to a targeted mean tidal volume of 6 to 8 ml/kg; the maximal inspiratory pressure ≤40 cmH2O; the flow trigger is set at 2 l/min; inspiratory cycling-off at 25% of peak flow; PEEP and FiO2 for oxygen saturation SaO2 ≥92%, with PEEP ≥5 cmH2O.
  In patients ventilated with variable PSV, the pressure support variability is as high as possible (up to 100%), while not exceeding the maximal inspiratory pressure determined by the treating physician.
  Arms: Variable PSV
Device: Conventional PSV — Pressure support is to a targeted mean tidal volume of 6 to 8 ml/kg; the maximal inspiratory pressure ≤40 cmH2O; the flow trigger is set at 2 l/min; inspiratory cycling-off at 25% of peak flow; PEEP and FiO2 for oxygen saturation SaO2 ≥92%, with PEEP ≥5 cmH2O. The adjustment of pressure support until extubation follows these rules for both non-variable and variable PSV groups: pressure support is gradually adjusted in decrements (or increments) of 0 to 5 cmH2O. PEEP is decreased in steps of 0 to 5 cmH2O; PEEP and FiO2 are adjusted to achieve a SaO2 ≥92%, with a PEEP ≥5 cmH2O.
  Arms: Conventional PSV
Device: Automated PSV — Pressure support is to a targeted mean tidal volume of 6 to 8 ml/kg; the maximal inspiratory pressure ≤40 cmH2O; the flow trigger is set at 2 l/min; inspiratory cycling-off at 25% of peak flow; PEEP and FiO2 for oxygen saturation SaO2 ≥92%, with PEEP ≥5 cmH2O.Smart CareTM as total automated procedure will be used.
  Arms: Automated PSV
Device: NAVA — NAVA level is to a targeted mean tidal volume of 6 to 8 ml/kg; the maximal inspiratory pressure ≤40 cmH2O; the Edi level was increased by step of 0,2 cm/h2o/ mcvolt, PEEP and FiO2 for oxygen saturation SaO2 ≥92%, with PEEP ≥5 cmH2O.
  Arms: NAVA

SUMMARY:
The aim of this multicenter, randomized controlled trial is to evaluate the weaning time from mechanical ventilation comparing non-variable PSV, variable PSV, and Smart CareTM.

This study is a multicenter randomized controlled open trial comparing variable, non-variable pressure support ventilation and Smart CareTM in patients receiving mechanical ventilation for more than 24 hours who are able to be weaned.

The aim of the study is to determine the duration of weaning from mechanical ventilation for each one of the above mentioned weaning methods

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* duration of controlled mechanical ventilation≥ 24 h
* temperature≤ 39°C
* hemoglobin≥ 6 g/dl
* ratio of arterial partial pressure of oxygen to inspiratory oxygen fraction - PaO2/FiO2≥150mmHg with positive end-expiratory pressure (PEEP)≤ 16 cmH2O
* ability of the patient to breathe spontaneously
* informed consent

Exclusion Criteria:

* patient participated in another interventional trial within the last four weeks before enrollment
* peripheral neurological disease associated with impairment of the respiratory pump
* muscular disease associated with impairment of the respiratory pump
* unstable thorax with paradoxical chest wall movement
* planned surgery under general anesthesia within 72 hours
* difficult airway or intubation
* existing tracheotomy at ICU admission
* expected survival<72 hours
* home mechanical ventilation or on chronic oxygen therapy
* suspected or confirmed pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
weaning time | within 6 hours
  weaning time defined as the time from randomization to successful extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: No